CLINICAL TRIAL: NCT06682429
Title: Telerehabilitation In The Home After Stroke: A Randomized, Controlled, Assessor-Blind Clinical Trial
Brief Title: Telerehabilitation In The Home After Stroke
Acronym: TR-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Moss Rehabilitation Research Institute (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, FAAN, FAHA, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Q221354
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; telehealth
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Patients are randomized to TR + usual care or usual care alone
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants in the usual care group will receive no TR, but will continue with the recommendations made by their care team. All participants in this group will be offered TR at the end of the study.
- Telerehabilitation + Usual Care (Experimental): Patients will receive 36 telerehabilitation sessions targeting arm motor function in addition to their usual care. TR consists of 70 minutes/day of activities targeting arm function, 6 days/week for 6 weeks. Half of these sessions are supervised by a licensed therapist, and the other half are done independently.
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. TR sessions will be a combination of games, exercises, stroke education, assessments, in addition to videoconferencing with therapists to discuss progress, issues, goals, and changes to the treatment plan.
  Arms: Telerehabilitation + Usual Care

SUMMARY:
The purpose of this research study is to evaluate whether telerehabilitation targeting arm movement, when added to usual care, improves arm function and reduces global disability after stroke, compared to usual care alone.

Patients with arm weakness due to stroke that happened in the past 90-150 days will be randomized into one of two groups: [1] TR and usual care; [2] usual care only (no TR), but people in the usual care group will be offered TR once the study is done. TR consists of 70 minutes/day of activities targeting arm function, 6 days a week for 6 weeks.

DETAILED DESCRIPTION:
This is a randomized, assessor-blinded study that involves the use of telerehabilitation to deliver additional therapy for persons with stroke. Patients with arm weakness due to stroke that happened in the past 90-150 days will be randomized into one of two groups: [1] TR and usual care; [2] usual care only (no TR), but people in the usual care group will be offered TR once the study is done. TR consists of 70 minutes/day of activities targeting arm function, 6 days a week 6-8 weeks. The hypothesis of this study is patients receiving TR in addition to their usual care will have significantly greater recovery of arm function compared to patients receiving usual care alone.

Study participation will last approximately 8 months and includes 4 in-person visits. At these visits, patients will undergo a variety of assessments including tests of arm function and a single MRI scan of the brain. Patients undergoing TR will receive arm motor training, which consists of 36 sessions of assigned exercises, games, and stroke education; these total 70 minutes in length and occur 6 days a week for 6 weeks; TR subjects will also continue usual care. Patients in the usual care group only will not engage in TR but will instead continue all of the therapies recommended by their medical team. At the end of the study, participants in the usual care group will be offered TR.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years at the time of randomization
2. The index stroke was radiologically verified, due to ischemia or intracerebral hemorrhage (ICH), and had time of onset 120±30 days prior to randomization
3. The stroke caused upper extremity deficits as defined by Action Research Arm Test score 18-44 (out of 57) at Baseline Visit 1
4. Box & Block Test score with affected arm is ≥1 block in 60 seconds at Baseline Visit 1
5. Able to successfully perform all 3 rehabilitation exercise test examples (simple commands) at Baseline Visit 1
6. Informed consent and behavioral contract signed by the subject (i.e., no surrogate consent)

Exclusion Criteria:

1. A major, active, coexistent neurological, psychiatric, or medical disease that reduces the likelihood that a subject will be able to comply with all study procedures
2. Unable or unwilling to perform study procedures/therapy, or expectation of noncompliance with study procedures/therapy, or expectation that subject cannot participate in all study visits
3. A diagnosis (apart from the index stroke) that substantially affects paretic arm function
4. Severe depression, defined as Geriatric Depression Scale Score >10/15 at Baseline Visit 1
5. Significant cognitive impairment, defined as Montreal Cognitive Assessment score <22 [a lower score is permitted if due to aphasia and allowed by the site PI]
6. Deficits in communication that interfere with reasonable study participation
7. Severe UE spasticity, defined as presence of contracture or modified Ashworth Scale score=4 in either biceps or pectoralis
8. Modified Rankin Scale score was >2 prior to the index stroke
9. A new symptomatic stroke has occurred since the index stroke, or a separate stroke occurred within 30 days prior to the index stroke
10. Lacking visual acuity, with or without corrective lens, of 20/50 or better in at least one eye
11. Life expectancy < 9 months
12. Pregnant; women of child-bearing potential must have a negative pregnancy test
13. Botulinum toxin to the paretic arm: received in the prior 3 months OR expected by the 8-Month Visit
14. Concurrent enrollment in another therapy-based investigational study where the duration of the investigational therapy's activity is likely to occur during the subject's participation in the study
15. Subject lacks sufficient English or Spanish to comply with study procedures and TR instructions
16. Expectation that subject will not have a single domicile address during the 6 weeks of therapy that is within 1.5-hr drive of the central study site [this can be waived at the discretion of the site PI]
17. Contraindication to MRI
18. On isolation precautions, e.g., due to active COVID-19

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in Action Research Arm Test (ARAT) Score from Baseline to 2 Months | 2 months
  The ARAT scale measures arm function using a scale that runs from 0 to 57 points, with higher numbers reflecting better arm function.

SECONDARY OUTCOMES:
Change in modified Rankin Scale (mRS) Score from Baseline to 2 Months | 2 months
  The mRS scale measures global function using a scale that runs from 0 to 6 points, with lower numbers reflecting better global function.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cramer, MD, Principal Investigator — University of California, Los Angeles
Locations (19):
- United States (19):
  - Rancho Los Amigos Research Institute, Downey, California
  - Keck Medical Center of USC, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Casa Colina Hospital and Centers for Healthcare, Pomona, California
  - Hillcrest Medical Center at UC San Diego Health, San Diego, California
  - Brooks Rehabilitation Hospital, Jacksonville, Florida
  - Emory Rehabilitation Hospital, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - NYP Columbia University Medical Center, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Jefferson Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UTHealth Houston - Institute for Stroke and Cerebrovascular Diseases, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Non-PHI data will be shared with appropriate parties after the study is completed and published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Any time after September 30, 2030
Access Criteria: Appropriate parties with appropriate intention for use of the data, starting 9/30/30, with access to PHI-free data.